CLINICAL TRIAL: NCT05126654
Title: Development of a Partially Hydrolyzed Guar Gum (PHGG) Based Synbiotic for Amelioration of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Partially Hydrolyzed Guar Gum (PHGG) for Amelioration of Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJUH110120
Record Dates: First submitted 2021-10-12; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: COPD; Microbial Colonization; Respiratory Tract Disease
Keywords: COPD; Gut microbiota; Respiratory tract; prebiotics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Communicable Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD with PHGG (Experimental): COPD patient PHGG 5g/day for 1 month
  Interventions: Dietary Supplement: Partially Hydrolyzed Guar Gum (PHGG)
- COPD without PHGG (No Intervention): COPD patient without PHGG 5g/day for 1 month
- Healthy with PHGG (Active Comparator): Healthy PHGG 5g/day for 1 month
  Interventions: Dietary Supplement: Partially Hydrolyzed Guar Gum (PHGG)
- Healthy without PHGG (No Intervention): Healthy without PHGG 5g/day for 1 month

INTERVENTIONS:
Dietary Supplement: Partially Hydrolyzed Guar Gum (PHGG) — Partially Hydrolyzed Guar Gum 5 gram/day for 1 month
  Arms: COPD with PHGG; Healthy with PHGG

SUMMARY:
Some components of the diet could promote the growth of certain bacterial strains present in the intestine, which are closely associated with benefits for host health. An intestinal commensal Parabacteroides goldsteinii (Pg) was highlighted to be significantly negatively associated with severity of COPD. Furthermore, the investigators identify the potential prebiotics (PHGG) which may enrich the abundance of P. goldsteinii and increase the probiotic effect of P. goldsteinii.

The investigators designed a randomized control study, which enroll adults diagnosed with COPD. Then the two groups will receive PHGG or not. Stool samples will be collected. The ameliorative efficacy will be evaluated by questionnaire and lung function test. Intestinal microbiota and metabolome will be analyzed and the correlation with lung function indices will be further investigated.

DETAILED DESCRIPTION:
It is well known that some components of the diet could promote the growth of certain bacterial strains present in the intestine, which are closely associated with benefits for host health. In the previous study, the investigators found that an intestinal commensal Parabacteroides goldsteinii (Pg) was highlighted to be significantly negatively associated with severity of COPD. Furthermore, the investigators identify the potential prebiotics (PHGG) which may enrich the abundance of P. goldsteinii and increase the probiotic effect of P. goldsteinii. However, the effect of PHGG supplement on compositional and functional properties of the human microbiota with COPD still remains unclear.

In this proposal, the investigators designed a randomized control study, which enroll adults diagnosed with COPD. The investigators will review their past medical records and related image and lung function test. Then the two groups will receive PHGG or not. Stool samples will be collected. The ameliorative efficacy will be evaluated by questionnaire and lung function test. Intestinal microbiota and metabolome will be analyzed and the correlation with lung function indices will be further investigated. In the future, it may be used to investigate and analyze the change of microbiota and metabolome, then develop possible treatment options of COPD.

ELIGIBILITY:
Inclusion Criteria:

* age of 40-85 years
* diagnosis of COPD made by pulmonologist
* provision of written informed consent

Exclusion Criteria:

* severe and unstable comorbidities or active malignancy
* COPD exacerbation within the 4 weeks prior
* cognitive impairment or a psychiatric disorder
* pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale (mMRC) | after PHGG 5 gram/day for 1 month
  change of mMRC scale, 0 the best, 4 the worst
COPD Assessment Test (CAT) | after PHGG 5 gram/day for 1 month
  change of CAT (0 the best, 40 the worst)
St. George's Respiratory Questionnaire (SGRQ) | after PHGG 5 gram/day for 1 month
  change of SGRQ score, 0 the best, 100 the worst
FEV1 | after PHGG 5 gram/day for 1 month
  change of FEV1
FEV1% | after PHGG 5 gram/day for 1 month
  change of FEV1%
FVC | after PHGG 5 gram/day for 1 month
  change of FVC
FVC% | after PHGG 5 gram/day for 1 month
  change of FVC%
FEV1/FVC% | after PHGG 5 gram/day for 1 month
  change of FEV1/FVC%
FEV3 | after PHGG 5 gram/day for 1 month
  change of FEV3
FEV3% | after PHGG 5 gram/day for 1 month
  change of FEV3%
FEV3/FVC% | after PHGG 5 gram/day for 1 month
  change of FEV3/FVC%
MMEF | after PHGG 5 gram/day for 1 month
  change of MMEF
MMEF% | after PHGG 5 gram/day for 1 month
  change of MMEF%
PEF | after PHGG 5 gram/day for 1 month
  change of PEF
PEF% | after PHGG 5 gram/day for 1 month
  change of PEF%
blood cytokine | after PHGG 5 gram/day for 1 month
  change of blood cytokine
Microbiota of stool | after PHGG 5 gram/day for 1 month
  change of stool microbiota contribution

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chen Lu, PhD, Principal Investigator — Department of Respiratory Therapy, College of Medicine, Fu-Jen Catholic University, Taiwan
Locations (1):
- Yen-Liang Kuo, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No